CLINICAL TRIAL: NCT03662139
Title: Reliability and Validity of the Dynamic Gait Index in Children With Hemiplegic Cerebral Palsy
Brief Title: Dynamic Gait Index in Hemiplegic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 02.04.2018-113
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2019-11-05 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-11

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy; Gait Disorders, Neurologic
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Palsy Group: 16 patients will be included. Dynamic Gait Index and other assessments will be performed twice with a 7 - 10 day interval by two evaluators
  Interventions: Other: Dynamic Gait Index
- Healthy Control Group: 16 healthy children will be included. Dynamic Gait Index and other assessments will be performed twice with a 7 - 10 day interval by two evaluators
  Interventions: Other: Dynamic Gait Index

INTERVENTIONS:
Other: Dynamic Gait Index — Dynamic Gait Index is a clinical tool for assessing functional balance and gait variability in people with neurologic conditions

SUMMARY:
The purpose of this study is to assess validity and reliability of Dynamic Gait Index (DGI) in patients with unilateral spastic cerebral palsy

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a childhood onset, lifelong neurological disorder, attributed to non-progressive injury of the fetal or immature brain. It causes movement deterioration and activity limitation. In CP patients increase in slow walking speed, shorter step length, and longer duration in the double support phase are common. Such gait changes are thought to reflect the unbalanced walking pattern seen in these children. Although children with CP are well known to have poor balance and high fall incidence, little effort has been made to quantify the dynamic walking stability of these children.

The Dynamic Gait Index (DGI) is a performance-based tool developed by Shumway-Cook and Woollacott to quantitatively measure dynamic balance capabilities. It also evaluates the individual's ability to modify gait in response to changing gait task requirements. Despite it's widespread use in the elderly population, DGI has not yet been investigated in children with neurological conditions. Considering that it takes a little time to apply the test, it may be advantageous for children in terms of simplicity and ease of administration.

In this study the investigators aim to validate and assess interrater and test - retest reliabilities of Turkish version of Dynamic Gait Index in children with unilateral, spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spastic unilateral cerebral palsy
* Age between 4 - 16
* Able to stand and walk without any orthosis or special equipment
* Volunteer to study

Exclusion Criteria:

* Being unable to walk
* Having cognitive disorder
* History of orthopedic surgery or any intervention for spasticity within the previous 12 months
* Uncontrolled epilepsy
* Visual conditions that prevent full participation to assessments
* Lower extremity contracture that may affect assessments

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 16 spastic unilateral cerebral palsy patients, between 6 - 14 years of age, and 16 healthy volunteer peers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag Saygi, Prof, Study Chair — Department of PM&R, Marmara University School of Medicine; Ayca Evkaya, PT, Principal Investigator — Department of PM&R, Marmara University School of Medicine
Locations (1):
- Marmara University School of Medicine, Pendik Research and Education Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Shumway-Cook A, Taylor CS, Matsuda PN, Studer MT, Whetten BK. Expanding the scoring system for the Dynamic Gait Index. Phys Ther. 2013 Nov;93(11):1493-506. doi: 10.2522/ptj.20130035. Epub 2013 Jun 27. PMID 23813090
- [Background] Bandong AN, Madriaga GO, Gorgon EJ. Reliability and validity of the Four Square Step Test in children with cerebral palsy and Down syndrome. Res Dev Disabil. 2015 Dec;47:39-47. doi: 10.1016/j.ridd.2015.08.012. Epub 2015 Aug 27. PMID 26318393
- [Background] Carey H, Martin K, Combs-Miller S, Heathcock JC. Reliability and Responsiveness of the Timed Up and Go Test in Children With Cerebral Palsy. Pediatr Phys Ther. 2016 winter;28(4):401-8. doi: 10.1097/PEP.0000000000000301. PMID 27661230
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Derived] Evkaya A, Karadag-Saygi E, Karali Bingul D, Giray E. Validity and reliability of the Dynamic Gait Index in children with hemiplegic cerebral palsy. Gait Posture. 2020 Jan;75:28-33. doi: 10.1016/j.gaitpost.2019.09.024. Epub 2019 Sep 23. PMID 31590067

RESULTS

PARTICIPANT FLOW:
Groups:
- Cerebral Palsy Group: 16 patients with hemiplegic cerebral palsy will be included. Dynamic Gait Index and other assessments will be performed twice with a 7 - 10 day interval by two evaluators
  Dynamic Gait Index: Dynamic Gait Index is a clinical tool for assessing functional balance and gait variability in people with neurologic conditions
Period: Overall Study
Arm/Group | Cerebral Palsy Group | Healthy Control Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cerebral Palsy Group | Healthy Control Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.31 (2.62) | 9.75 (2.51) | 10.03 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 11 | 8 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 142 (15) | 140 (13) | 141 (14)
Body weight [Mean (Standard Deviation); unit: kg] | 38.43 (10.85) | 38.87 (11.63) | 38.65 (11.07)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.56 (3.12) | 19.40 (3.23) | 18.98 (3.16)
Gestational week [Mean (Standard Deviation); unit: weeks] | 35.12 (4.22) | 37.25 (2.38) | 36.19 (3.54)
Birth weight (kg) [Mean (Standard Deviation); unit: kg] | 2.52 (0.78) | 3.03 (0.67) | 2.77 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Gait Index (DGI)
Description: Dynamic Gait Index is a tool consisting eight items; gait on a flat surface, changing speed, gait with horizontal and vertical head turns, pivot turn, stepping over obstacle, Minimum score is 0, maximum score is 24, higher scores indicate better outcome. Scores lower than 19 indicate risk of falling and above 22 define safe ambulance.
Time Frame: Day 1 (Baseline) in both groups (Cerebral Palsy group same day by two different evaluators), Day 7-10 in the Cerebral Palsy group only
Population: Cerebral palsy group is assessed 2 times in a 7-10 days period for the test-retest reliability. Control group is assessed only once.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cerebral Palsy Group | Healthy Control Group
Number analyzed (Participants) | 16 | 16
units on a scale
  1. Assessment | 19 [8 to 23] | 24 [23 to 24]
  2. Assessment: number analyzed (Participants) | 16 | 0
  2. Assessment | 18.5 [10 to 23] |
Statistical Analysis 1: Comparison: Cerebral Palsy Group vs Healthy Control Group; Between group difference; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cerebral Palsy Group; Test - Retest Reliability (Difference between 1st and 2nd assessments in Cerebral Palsy group); Test type: Superiority; p < 0.05, Intraclass Correlation Coefficient(ICC); Two-way random-effect model; ICC = 0.97, 95% CI 2-sided [0.915 to 0.99] — Reliability estimates were interpreted as follows: >0.90=excellent; 0.75-0.90=good; 0.50-0.75=medium; <0.50=low
Statistical Analysis 3: Comparison: Cerebral Palsy Group; Interrater Reliability (Difference between 1st and 2nd evaluators in Cerebral Palsy group); Test type: Superiority; p < 0.01, Intraclass Correlation Coefficient(ICC); Two-way random-effect model; ICC = 0.983, 95% CI 2-sided [0.882 to 0.998] — Reliability estimates were interpreted as follows: >0.90=excellent; 0.75-0.90=good; 0.50-0.75=medium; <0.50=low

2. Secondary Outcome: Pediatric Balance Scale (PBS)
Description: Pediatric Balance Scale is a functional balance scale adapted and customized from Berg Balance Scale for use with children. Pediatric Balance Scale is a 14-item, criterion-referenced measure, which examines functional balance in the context of everyday tasks. It can easily be administered and scored in less than 20 minutes using equipment commonly found in schools and clinics. Scoring (0-4) is based on how long a specific movement or position is performed, how long the position can be maintained, or how much assistance it requires. Minimum score is 0, maximum score is 56; higher scores indicate better dynamic balance.
Time Frame: Only Day 1 in both Cerebral Palsy and Healthy control groups (Cerebral Palsy group same day by two different evaluators)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cerebral Palsy Group | Healthy Control Group
Number analyzed (Participants) | 16 | 16
units on a scale
  1. Assessment | 49.5 [39 to 54] | 56 [53 to 56]
  2. Assessment: number analyzed (Participants) | 16 | 0
  2. Assessment | 50 [39 to 54] |
Statistical Analysis 1: Comparison: Cerebral Palsy Group vs Healthy Control Group; Between group difference; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cerebral Palsy Group; Correlation between Dynamic Gait Index (DGI) and Pediatric Balance Scale (PBS) scores in Cerebral Palsy group; Test type: Superiority; p < 0.05, Spearman's Correlation Test; The level of relationship was classified as follows <0.30=small/negligible; 0.30-0.50=low; 0.50-0.70=moderate; 0.70-0.90=high; >0.90=very high; Spearman's correlation coefficient (rs) = 0.724

3. Secondary Outcome: Timed Up and Go Test (TUG)
Description: TUG is a test determining fall risk and balance by their physical performance in sitting to standing, and walking. Test begins with the patient sitting back in a standart chair and when asked walking 10 feets on a certain line than back to the chair sitting. Completion time is recorded for the task and longer time indicates worse ambulation and higher risk of fall.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | Cerebral Palsy Group | Healthy Control Group
Number analyzed (Participants) | 16 | 16
seconds
  1. Assessment | 10 [5.87 to 16.22] | 6.97 [5.15 to 8.42]
  2. Assessment: number analyzed (Participants) | 16 | 0
  2. Assessment | 8.72 [6.16 to 14.23] |
Statistical Analysis 1: Comparison: Cerebral Palsy Group vs Healthy Control Group; Between group difference; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cerebral Palsy Group; Correlation between Dynamic Gait Index (DGI) and Timed Up and Go Test (TUG) scores in Cerebral Palsy group; Test type: Superiority; p < 0.01, Spearman's Correlation Test; Spearman's correlation coefficient (rs) = -0.828 — The level of relationship was classified as follows <0.30=small/negligible; 0.30-0.50=low; 0.50-0.70=moderate; 0.70-0.90=high; >0.90=very high

4. Secondary Outcome: Four Square Step Test (FSST)
Description: FSST, assesses dynamic balance and coordination through stepping forwards, sideways, and backwards in a timed fashion. It is a valid and reliable tool in children with cerebral palsy. The test requires the participant to step forwards, backwards and sideways over four-square shaped line in a specified sequence. Completion time is recorded for the task and longer time indicates worse ambulation and higher risk of fall.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | Cerebral Palsy Group | Healthy Control Group
Number analyzed (Participants) | 16 | 16
seconds
  1. Assessment | 11.85 [8.35 to 40.38] | 7.33 [6.25 to 10.20]
  2. Assessment: number analyzed (Participants) | 16 | 0
  2. Assessment | 10.21 [7.42 to 38.42] |
Statistical Analysis 1: Comparison: Cerebral Palsy Group vs Healthy Control Group; Between group difference; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cerebral Palsy Group; Correlation between Dynamic Gait Index (DGI) and Four Square Step Test (FSST) scores in Cerebral Palsy group; Test type: Superiority; p < 0.05, Spearman's Correlation Test; Spearman's correlation coefficient (rs) = -0.673 — [estimate comment as in outcome 3, analysis 2]

ADVERSE EVENTS:
Time Frame: 7 - 10 days
Groups:
- Cerebral Palsy Group: 16 patients with hemiplegic cerebral palsy will be included. Dynamic Gait Index and other balance assessments will be performed twice with a 7 - 10 day interval by two evaluators
- Healthy Control Group: 16 healthy children will be included. Dynamic Gait Index and other balance assessments will be performed twice with a 7 - 10 day interval by two evaluators
Arm/Group | Cerebral Palsy Group | Healthy Control Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03662139/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03662139/SAP_001.pdf